CLINICAL TRIAL: NCT00846469
Title: 64 Slice Coronary CT Angiography vs. Standard Therapy in the Emergency Room: Determining Cost-effectiveness and Predicting Clinical Outcome in Patients With Low and Moderate Risk for Acute Coronary Syndrome.
Brief Title: Coronary Computed Tomography (CT) Angiography Versus Standard Therapy in the Emergency Room
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Suzanne Chong, MD, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM 0000 7282
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Chest Pain
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- chest pain (Experimental): CCTA (Coronary computed tomography angiography)
  Interventions: Procedure: CCTA (coronary computed tomography angiography); Other: Control section

INTERVENTIONS:
Procedure: CCTA (coronary computed tomography angiography) — A CCTA (coronary computed tomography angiography) scan is a CT scan of the blood vessels of the heart. This CCTA (Coronary Computed Tomography Angiography)will be performed and a contrast medication will be injected through an IV line to help make the CT pictures more clear. Medication may or may not be given to control your heart rate during the scan. After the scan is completed it will be read. Your emergency room physician will use the CT results to determine your treatment.
Other: Control section — Normal emergency room treatment for symptoms of chest pain.

SUMMARY:
The purpose of this study is to determine the usefulness of CCTA (Coronary Computed Tomography Angiography) in the emergency room setting to diagnose and predict the outcome of patients with chest pain who have a low to moderate risk of heart disease.

And to also determine if the use of CCTA(Coronary Computed Tomography Angiography) is more cost effective (cost less) than the current standards of care treatments. To determine if patients who present to the emergency room w/low to moderate probability of having an ACS (Acute Coronary Syndrome) prefer CCTA (coronary computed tomography angiography)-based care compared to standard algorithm based care.

ELIGIBILITY:
Inclusion Criteria:

* 25 years of age or older
* Experiencing chest pain

Exclusion Criteria:

* Pregnant
* At high risk for ACS (Acute Coronary Syndrome)

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To assess the usefulness of CCTA (coronary computed tomography angiography)in the emergency room setting to diagnose/predict the outcome of patients w/chest pain who have low to moderate risk of heart disease. | one year

SECONDARY OUTCOMES:
To determine if the use of CCTA (coronary computed tomography angiography)is more cost effective than the current standard of care treatments being used. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Chong, MD, Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States